CLINICAL TRIAL: NCT00048477
Title: Determination of Nitrite as a Source of Bioactive Nitric Oxide in Human Subjects
Brief Title: Effects of Nitrite on Blood Vessel Dilation in Normal Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030020; 03-H-0020
Record Dates: First submitted 2002-10-31; First posted 2002-11-01 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-11

CONDITIONS: Nitric Oxide; Endothelium-Derived Relaxing Factor; Healthy
Keywords: Endothelium; Vasodilation; Exercise; Hemoglobin; Blood Flow; Healthy Volunteer; HV
MeSH Terms: conditions — Aneurysm; Motor Activity | interventions — omega-N-Methylarginine; Sodium Nitrite

INTERVENTIONS:
Drug: L-NMMA and Sodium Nitrite

SUMMARY:
Nitric oxide gas is important in regulating blood vessel dilation, and consequently, blood flow. This gas is continuously produced by endothelial cells, which line the blood vessels. This study will examine whether nitrite, a molecule that normally circulates in the blood stream, can also dilate blood vessels. The results of this study may be valuable in developing treatments for people with conditions associated with impaired endothelial production of nitric oxide, including high blood pressure, high blood cholesterol, diabetes, estrogen deficiency, and others.

Healthy, non-smoking normal volunteers 21 years of age or older may be eligible for this study. People who lack the enzyme G6PD or cytochrome B5 in their red blood cells may not participate. Absence of these enzymes can lead to episodes of sudden shortness of breath and cyanosis (blueness of the skin due to lack of sufficient oxygen). Participants will undergo the procedures described in study Parts A and B, as follows:

* Part A - After numbing the skin, small tubes are placed in the artery and vein at the inside of the elbow of the dominant arm (right- or left-handed) and a small tube is placed in a vein of the other arm. The tubes are used for infusing saline (salt water) and for drawing blood samples. A pressure cuff is placed around the upper part of the dominant arm, and a rubber band device called a strain gauge is also placed around the arm to measure blood flow. When the cuff is inflated, blood flows into the arm, stretching the strain gauge at a rate proportional to the flow. Grip-strength of the dominant arm is measured with a dynamometer to determine maximum grip-strength. Then, several measurements of blood flow, nitrite, hemoglobin, and handgrip are made before and after administration of L-NMMA, a drug that blocks endothelial production of nitric oxide.
* Part B - Part A testing is repeated, except that sodium nitrite dissolved in a saline solution is infused into the artery of the forearm for a few minutes before and during the hand-grip exercises. In addition, blood samples are drawn before and after each handgrip exercise to measure methemoglobin, a substance that, at excessive levels, can cause adverse side effects.

DETAILED DESCRIPTION:
Nitric oxide (NO) is a soluble gas continuously synthesized by the endothelium and contributes importantly to vasodilator tone of the coronary and systemic circulations by activating guanylyl cyclase in vascular smooth muscle, causing relaxation. Although regional synthesis of NO by the endothelium contributes to local vasodilator tone, we have shown previously that NO may be transported in blood, and have biological effects at a distance from the site of entry into the circulation. Thus, we found that NO may be transported bound to heme iron in red blood cells and released at vascular sites of deficient NO synthesis, restoring vasodilator tone. Another potential source of bioactive NO is via nitrite, formed by the auto-oxidation of NO. This study is designed to determine the contribution of nitrite transported in blood to forearm microvascular dilator tone in healthy subjects at rest and during regional hypoxia associated with forearm exercise stress, with measurements made before and after regional blockade of endothelial NO synthesis. Findings in this study may be relevant to understanding the physiological contribution and therapeutic potential of nitrite in the regulation of vasodilator tone in diseases and conditions associated with regional endothelial dysfunction and reduced endothelial NO bioactivity (e.g., hypertension, diabetes mellitus, hypercholesterolemia, cigarette smoking, estrogen deficiency).

ELIGIBILITY:
INCLUSION CRITERIA

All volunteer subjects must be at least 21 years of age in good health and have provided informed, written consent for participation in this study.

EXCLUSION CRITERIA

Subjects with a history or evidence of present or past hypertension (blood pressure greater than 145/95 mmHg), hypercholesterolemia (LDL cholesterol greater than 130 mg/dL), diabetes mellitus (fasting blood glucose greater than 130 mg/dL), smoking within two years, cardiovascular disease, peripheral vascular disease, coagulopathy, or any other disease predisposing to vasculitis or Raynaud's phenomenon.

All subjects will be tested for red blood cell G6PD deficiency; levels below the lower limits of normal will result in exclusion from participation in the study.

Subjects with a known cytochrome B5 deficiency will not participate in this study.

Subjects with a history of reaction to a medication or other substance characterized by dyspnea and cyanosis will not participate in this study.

Subjects with a baseline methemoglobin level greater than 1% will not receive nitrite infusions.

Lactating and pregnant females.

No volunteer subject will be allowed to take any medication (oral contraceptive agents are allowed), vitamin supplements, herbal preparations, nutriceuticals or other 'alternative therapies' for at least one month prior to study and will not be allowed to take aspirin for one week prior to study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Start 2002-10; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Background] Palmer RM, Ferrige AG, Moncada S. Nitric oxide release accounts for the biological activity of endothelium-derived relaxing factor. Nature. 1987 Jun 11-17;327(6122):524-6. doi: 10.1038/327524a0. PMID 3495737
- [Background] Palmer RM, Ashton DS, Moncada S. Vascular endothelial cells synthesize nitric oxide from L-arginine. Nature. 1988 Jun 16;333(6174):664-6. doi: 10.1038/333664a0. PMID 3131684